CLINICAL TRIAL: NCT01973738
Title: Comparison of the Clinical Efficacy and Safety Between Raloxifene and Bazedoxifene in Postmenopausal Women.
Brief Title: Comparison Between Raloxifene and Bazedoxifene
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Toshihiko Kono (Other)
Responsible Party: Sponsor-Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Organization: Tomidahama Hospital (Other)
Other Study IDs: IRB TH 05
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Selective Estrogen Receptor Modulator
Keywords: raloxifene; bazedoxifene; bone mineral density; bone turnover markers; bone quality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although there are two kinds of selective estrogen receptor modulator (SERM) :raloxifene (RLX) and bazedoxifene (BZA), the difference is still unclear. In this study, we plan to compare clinical efficacy and safety between RLX and BZA.

DETAILED DESCRIPTION:
Selective estrogen receptor modulator (SERM) is an important option for postmenopausal osteoporosis. There are two SERM approved in Japan for the treatment of postmenopausal osteoporosis in women at increased risk of fracture. One is raloxifene (RLX), and the other is bazedoxifene (BZA). There are few reports concerning to the clinical efficacy and safety data. In this study, we plan to compare clinical efficacy and safety between RLX and BZA.

The main objective of this study is to reveal the effects of RLX and BZA on bone mineral density, bone turnover markers, and bone quality markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women

Exclusion Criteria:

* Patients who could not use SERM

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporosis patients using SERM more for five years.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Effects of raloxifene vs. bazedoxifene on bone mineral density, bone turnover markers and bone quality markers in postmenopausal osteoporosis. | Up to 72 months
  The investigators plan to analyze 300 patients who undergo selective estrogen receptor modulator (SERM) treatments for five years.
  We investigate the efficacy of two SERMs: raloxifene (RLX) and bazedoxifene (BZA). Bone mineral density (BMD) andd laboratory analyses (bone markers, routine chemistry, urine, and bone quality marker of pentosidine) at baseline and every four to six months. We also investigate the side effects. Statical analyses are performed using Spearman correlation coefficients, paired t-test, Mann-Whitney U test, chi-square test and Fisher's exact test to compare the efficacy and safy between RLX and BZA.

CONTACTS AND LOCATIONS:
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan